CLINICAL TRIAL: NCT03992937
Title: Vaginal Micronized Progesterone or Levonorgestrel-releasing Intrauterine System (LNG-IUS) for Treatment of Non-atypical Endometrial Hyperplasia: A Prospective Randomized Trial
Brief Title: Vaginal Micronized Progesterone Versus Levonorgestrel for Treatment of Non-atypical Endometrial Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VMP vs LNG
Record Dates: First submitted 2019-06-14; First posted 2019-06-20 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Endometrial Hyperplasia Without Atypia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Micronized Progesterone (Experimental): Micronized progesterone tablets at a dose of 200 mg once a day vaginally, for 12 days (Between 14'th-25'th days of the menstrual cycle) over three months. With persistence of endometrial hyperplasia, the treatment is repeated for another 3 months
  Interventions: Drug: Vaginal Micronized Progesterone
- LNG-IUS (Active Comparator): Release rate of 20µg Levonorgestrel (Mirena-Intrauterine system) per day with one year follow up.
  Interventions: Device: Levonorgestrel-Intrauterine System

INTERVENTIONS:
Drug: Vaginal Micronized Progesterone — Micronized progesterone tablets at a dose of 200 mg once a day vaginally, for 12 days (Between 14'th-25'th days of the menstrual cycle) over three months.
  Arms: Vaginal Micronized Progesterone
Device: Levonorgestrel-Intrauterine System — Release rate of 20µg Levonorgestrel (Mirena-Intrauterine system) per day.
  Other Names: Mirena
  Arms: LNG-IUS

SUMMARY:
The purpose of this study is to compare the efficacy of the vaginal micronized progesterone and Levonorgestrel-releasing Intrauterine System for treatment of non-atypical endometrial hyperplasia in premenopausal women.

DETAILED DESCRIPTION:
Vaginal use of micronized progesterone in the treatment of endometrial hyperplasia can result in better than oral administration, as it will remain away from the first pass effect, and depending on the local application. In this study, we aimed to compare this local treatment with Levonorgestrel-releasing Intrauterine System for treatment of non-atypical endometrial hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Patients
* Patients with histologically confirmed endometrial hyperplasia without atypia

Exclusion Criteria:

* Endometrial hyperplasia with atypia
* Endometrial Carcinoma
* Suspected pathology on Physical/Ultrasonographic Examination e.g. fibroids, adnexal abnormality

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Regression and remission rate of endometrial hyperplasia | 3 month
  Endometrial sampling will be performed for 3'th month with Carmen canula. Pathological specimens will be reported by the specialist pathologist in accordance with the World Health Organisation (WHO) endometrial hyperplasia classification.

SECONDARY OUTCOMES:
Mean Reduction From Baseline in Menstrual Blood Loss | 6 month
  Menorrhagia Impact Questionnaire (MIQ). This is a validated disease-specific patient-reported outcome questionnaire assessing menstrual blood loss and the influence of heavy menstrual bleeding on quality of life
Number of Participants with adverse events associated with medication and device | 6 month
  Any side effects will be recorded into questionnaire during a consultation with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Şener Gezer, M.D, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tasci Y, Polat OG, Ozdogan S, Karcaaltincaba D, Seckin L, Erkaya S. Comparison of the efficacy of micronized progesterone and lynestrenol in treatment of simple endometrial hyperplasia without atypia. Arch Gynecol Obstet. 2014 Jul;290(1):83-6. doi: 10.1007/s00404-014-3161-4. Epub 2014 Feb 1. PMID 24488582
- [Derived] Gezer S, Kole E, Aksoy L. Vaginal micronized progesterone versus the levonorgestrel-releasing intrauterine system for treatment of non-atypical endometrial hyperplasia: A randomized controlled trial. Int J Gynaecol Obstet. 2023 May;161(2):661-666. doi: 10.1002/ijgo.14632. Epub 2023 Jan 12. PMID 36527262
- [Derived] Mittermeier T, Farrant C, Wise MR. Levonorgestrel-releasing intrauterine system for endometrial hyperplasia. Cochrane Database Syst Rev. 2020 Sep 6;9(9):CD012658. doi: 10.1002/14651858.CD012658.pub2. PMID 32909630